CLINICAL TRIAL: NCT02365662
Title: A Phase 1 Study of ABBV-221 in Subjects With Advanced Solid Tumor Types Likely to Exhibit Elevated Levels of Epidermal Growth Factor Receptor
Brief Title: A Study Evaluating Safety and Pharmacokinetics of ABBV-221 in Subjects With Advanced Solid Tumor Types Likely to Exhibit Elevated Levels of Epidermal Growth Factor Receptor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-429; 2014-003557-34 (EudraCT Number)
Record Dates: First submitted 2015-02-05; First posted 2015-02-19 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Non-small Cell Lung Cancer; Triple Negative Breast Cancer; Colorectal Carcinoma; Glioblastoma Multiforme
Keywords: Oncology; Cancer; Solid Tumor types likely to exhibit elevated levels of Epidermal Growth Factor Receptor; Solid Tumors
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Glioblastoma; Neoplasms | interventions — depatuxizumab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Solid Tumor Types Likely to Exhibit Elevated Levels of Epidermal Growth Factor Receptor
  Interventions: Drug: ABBV-221

INTERVENTIONS:
Drug: ABBV-221 — ABBV-221 will be given either every 3 weeks or 2 weeks on, 1 week off or weekly dosing by intravenous infusion approximately over 30 minutes to 3 hours. This is a dose escalation study, therefore the dose of ABBV-221 will change throughout the study.

SUMMARY:
This is an open-label, Phase I, dose escalation study to determine the recommended Phase 2 dose, maximum tolerated dose, and evaluate the safety and pharmacokinetic profile of ABBV-221 in participants with advanced solid tumors likely to exhibit elevated levels of Epidermal Growth Factor Receptor (EGFR).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 2.
* Has a solid tumor likely to exhibit elevated levels of EGFR (e.g. head and neck squamous cell carcinoma, non-small cell lung cancer, triple negative breast cancer ,colorectal carcinoma and glioblastoma multiforme).
* Has an archived, diagnostic tumor tissue available for analysis.
* Has adequate hematologic, renal, cardiac and hepatic function.
* Expanded Safety Cohort participants must have confirmed metastatic lung cancer and progressed after receiving prior platinum-containing chemotherapy.

Exclusion Criteria:

* Previously received an EGFR-directed monoclonal antibody within the past 4 weeks.
* Has unresolved, clinically significant toxicities from prior anti-cancer therapy defined as > Grade 1 on Common Terminology Criteria for Adverse Events.
* History of major immunologic reaction to any IgG containing agent.
* Any medical condition which in the opinion of the investigator places the participant at an unacceptably high risk for toxicities.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Measured for approximately 4 years
  Adverse event monitoring will be performed during the study
Maximum Plasma Concentration (Cmax) of ABBV-221 | Blood samples will be collected before infusion (0 hour, pre-dose) on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D5, C1D8, C1D15, C2D1, C3D1, C3D2, C3D3, C3D5, C3D8, C3D15, every 2 cycles starting with Cycle 5, and at the final visit (approximately 2 years).
  The maximum plasma concentration (Cmax; measured in ng/mL) is the highest concentration that a drug achieves in the plasma after administration in a dosing interval.
Area Under the Plasma Concentration-time Curve from 0 to the Time of the Last Measurable Concentration (AUCt) of ABBV-221 | Blood samples will be collected before infusion (0 hour, pre-dose) on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D5, C1D8, C1D15, C2D1, C3D1, C3D2, C3D3, C3D5, C3D8, C3D15, every 2 cycles starting with Cycle 5, and at the final visit (approximately 2 years).
  The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement of the total exposure of a drug in blood plasma.
Maximum tolerated dose of ABBV-221 | Up to 2 years from first dose of study drug.
  The highest dose level at which less than 2 of 6 participants or less than 33% of (if cohort is expanded beyond 6) participants experience a dose limiting toxicity.
Area Under the Plasma Concentration-time Curve of ABBV-221 | Blood samples will be collected before infusion (0 hour, pre-dose) on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D5, C1D8, C1D15, C2D1, C3D1, C3D2, C3D3, C3D5, C3D8, C3D15, every 2 cycles starting with Cycle 5, and at the final visit (approximately 2 years).
  The area under the plasma concentration-time curve (AUC; measured in ng*hr/mL) is a method of measurement of the total exposure of a drug in blood plasma.
Recommended Phase 2 dose of ABBV-221 | 1 day of study drug administration within the 21-day cycle at the designated cohort dose
  If a maximum tolerated dose (MTD) is reached, the recommended Phase 2 dose (RPTD) of ABBV-221 will not be a dose higher than the defined MTD, and will be selected based on the type(s) and occurrence(s) of dose limiting toxicities which occur in addition to the MTD. If a MTD is not reached, then the RPTD will be defined based on the safety and pharmacokinetic data.

SECONDARY OUTCOMES:
Assess the effect of systemic ABBV-221 administration on QT prolongation | At Days 1, 2, 3, 5, 8 of Cycle 1; Day 1 of every cycle starting at Cycle 2, and Final Visit (approximately 2 years from first dose of study drug)
  ECG parameters will be descriptively summarized, and the relationship between change of baseline of QT interval corrected for heart rate and concentration of three analytes will be explored.
Objective Response Rate (ORR) | At screening; at the end of Cycle 2 and the end of every 3 cycles for approximately 2 years from first dose of study drug
  ORR is the proportion of participants with objective response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (complete or partial objective response) will be calculated for all dosed participants with at least one measurable lesion at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (5):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Spain (2):
  - Fundacion Jimenez Diaz, Madrid
  - Hosp Univ Madrid Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Undecided